CLINICAL TRIAL: NCT02463903
Title: Coping Effectiveness Training in Patients With Chronic Heart Failure - a Randomized Controlled Trial
Brief Title: Coping Effectiveness Training in Patients With Chronic Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Swedish Red Cross University College (Other)
Responsible Party: Principal Investigator, Fredrik Saboonchi, Associate professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20140001
Record Dates: First submitted 2015-03-13; First posted 2015-06-04 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-06

CONDITIONS: Heart Failure
Keywords: Adaptation, Psychological; Heart Failure; Intervention Studies; Quality of Life; Hospital Readmission; Depression; Anxiety
MeSH Terms: conditions — Heart Failure; Depression; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Coping effectiveness Training (CET) (Experimental): The intervention consists of Coping Effectiveness Training (CET), a manual-based group intervention based on a cognitive transactional theory of stress and coping. The purpose of CET is to improve skills to appraise stress, teach a number of techniques to cope with stress, and to give an opportunity to interact with other people with similar experiences of living with CHF. The CET program will, in this study, be modified for patients with CHF. The intervention consists of seven, 90-minute weekly sessions led by a nurse with a Masters degree in nursing science and extensive experience in heart failure care in collaboration with a professional psychologist. Each group consisted of 8 to 12 patients.
  Interventions: Behavioral: Coping Effectiveness Training (CET)
- Control (No Intervention): The control group will receive standard health care and will not take part of the intervention.

INTERVENTIONS:
Behavioral: Coping Effectiveness Training (CET) — The participants in the intervention group will receive a work book explaining the theme and home assignment as well as providing a brief summary of every group session. The group leader has a manual. Both work book and manual have been translated to Swedish and adjusted to patients with chronic heart failure.
  Arms: Coping effectiveness Training (CET)

SUMMARY:
The purpose of the present study is to develop, implement and evaluate a stress management program aiming to improve emotional well-being, health-related quality of life and to reduce readmission to hospital in patients with chronic heart failure (CHF).

Method: A randomized controlled study design will be employed in which the intervention consists of Coping Effectiveness Training (CET), a manual-based group intervention based on a cognitive transactional theory of stress and coping. The purpose of CET is to improve skills to appraise stress, teach a number of techniques to cope with stress, and to give an opportunity to interact with other people with similar experiences of living with CHF. The control group will receive standard health care. The intervention group will receive seven weekly sessions of CET. Self-assessments of; emotional well-being, depression and anxiety, illness perception, health-related quality of life, coping strategies and social support will be performed before the intervention, directly after the intervention, six weeks, six months and one year after the intervention period as well as measuring readmission to hospital. In addition, the participants in the intervention group will fill in an anonymous written evaluation, with closed and open ended questions, directly after the intervention.

DETAILED DESCRIPTION:
Aim To develop, implement, and evaluate a stress management program, in form of patient education, to improve stress management and emotional well-being, health-related quality of life, as well as readmission to hospital in patients with chronic heart failure (CHF).

Hypothesis It is hypothesised that a Coping Effectiveness Training (CET) stress management program adapted for CHF improves stress management and emotional well-being (primary endpoint), health-related quality of life (secondary endpoint) and reduces readmission to hospital (tertiary endpoint) in patient with CHF.

Method A randomized controlled study design will be employed in which the intervention consists of patient education, Coping Effectiveness Training [CET]. CET is a manual based group intervention, which is based on the cognitive transactional theory of stress and coping. The CET programme will in this study be adjusted and modified to patients with CHF.

The control group (n=45) will receive standard health care. The intervention group (n=45) will receive CET intervention in form of patient education, led by a nurse with a master degree in nursing science and extensive experience in heart failure care. The intervention will consist of seven 90-minute weekly sessions. Each group will consist of 8 to 12 patients.

Measurements of the included variables will be performed before the intervention, directly after the intervention, six weeks, six months and one year after the intervention period. The following instruments will be employed for measuring outcome variables; PANAS for measuring emotional well-being; HADS for measuring depression and anxiety; B-IPQ for measuring the patients' appraisal and cognitive representation of of living with CHF; RAND-36 for measuring quality of life; Brief COPE for measuring coping strategies and thereby stress management and ESSI for measuring social support. Clinical variables that will be included are readmission to hospital and NYHA-class.

Data collection will be held at Danderyd Hospital. The inclusion criteria is patients diagnosed with CHF hospitalized at a heart failure ward or a heart failure outpatient clinic in Stockholm County Council, Sweden, are classified in NYHA-class II-III and are aged over 18 years. Exclusion criteria are cognitive dysfunction, life threatening disease such as cancer or primary organ failure and/or severe psychiatric diagnosis such as psychosis or severe depression, and not being able to understand the Swedish language.

Statistical analysis A preliminary power analysis, with a moderate effect size of Cohen's d = 0.50 and alpha = 0.05 indicates that to obtain a power of 0.80 a sample size of 90 patients (n=45 for each group) is needed (Cohen, 1988). MANOVA for repeated measurements for evaluating the intervention effect.

Readmission/health care consumption will be measured by:

1. Time to first readmission cardiovascular readmission or cardiovascular death.
2. Time to first readmission all cause or death despite cause.
3. Total time for inpatient care. Primary analysis will be conducted through MANCOVAS for repeated measures. Survival analysis (Kaplan Meyer and Cox regressions analysis) will be conducted for assessing the effect on readmissions to hospital.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with CHF hospitalized at a heart failure ward or a heart failure outpatient clinic in Stockholm County Council, Sweden, are classified in NYHA-class II-III and are aged over 18 years.

Exclusion Criteria:

* Cognitive dysfunction
* life threatening disease such as cancer or primary organ failure and/or severe psychiatric diagnosis such as psychosis or severe depression, and
* not being able to understand the Swedish language.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2011-03; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Emotional well-being (Composite measure of positive and negative affect) | Change from baseline to directly after, 6 weeks, 6 months and 1 year after intervention
  As measured by self-assessment questionnaire PANAS. Analysis will be conducted with Repeated measures ANCOVA.
Depression and anxiety (Composite measure) | Change from baseline to directly after, 6 weeks, 6 months and 1 year after intervention
  As measured by self-assessment questionnaire HADS. Analysis will be conducted with Repeated measures ANCOVA.

SECONDARY OUTCOMES:
Health-related quality of life (Composite measure) | Change from baseline directly after, 6 weeks, 6 months and 1 year after intervention
  As measured by self-assessment questionnaire RAND 36. Analysis will be conducted with Repeated measures ANCOVA.

OTHER OUTCOMES:
Readmission to hospital | During the entire follow-up period, mean follow-up time an average of 3 years (median) but at least 1 year. From start of the first intervention group to end of study-date.
  1. Time to first readmission cardiovascular readmission or cardiovascular death.
  2. Time to first readmission all cause or death despite cause.
  3. Total time for inpatient care.

CONTACTS AND LOCATIONS:
Overall Officials: Fredrik Saboonchi, Professor, Study Director — Swedish Red Cross University College

REFERENCES:
- [Background] Watson D, Clark LA, Tellegen A. Development and validation of brief measures of positive and negative affect: the PANAS scales. J Pers Soc Psychol. 1988 Jun;54(6):1063-70. doi: 10.1037//0022-3514.54.6.1063. PMID 3397865
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Background] Carver CS. You want to measure coping but your protocol's too long: consider the brief COPE. Int J Behav Med. 1997;4(1):92-100. doi: 10.1207/s15327558ijbm0401_6. PMID 16250744
- [Background] Broadbent E, Petrie KJ, Main J, Weinman J. The brief illness perception questionnaire. J Psychosom Res. 2006 Jun;60(6):631-7. doi: 10.1016/j.jpsychores.2005.10.020. PMID 16731240
- [Background] Berkman LF, Blumenthal J, Burg M, Carney RM, Catellier D, Cowan MJ, Czajkowski SM, DeBusk R, Hosking J, Jaffe A, Kaufmann PG, Mitchell P, Norman J, Powell LH, Raczynski JM, Schneiderman N; Enhancing Recovery in Coronary Heart Disease Patients Investigators (ENRICHD). Effects of treating depression and low perceived social support on clinical events after myocardial infarction: the Enhancing Recovery in Coronary Heart Disease Patients (ENRICHD) Randomized Trial. JAMA. 2003 Jun 18;289(23):3106-16. doi: 10.1001/jama.289.23.3106. PMID 12813116
- [Background] Hays RD, Sherbourne CD, Mazel RM. The RAND 36-Item Health Survey 1.0. Health Econ. 1993 Oct;2(3):217-27. doi: 10.1002/hec.4730020305. PMID 8275167
- [Background] Chesney MA, Folkman S. Psychological impact of HIV disease and implications for intervention. Psychiatr Clin North Am. 1994 Mar;17(1):163-82. PMID 8190663
- [Background] Lazarus, R.S., & Folkman, S. (1984). Stress, appraisal and coping. New York: Springer Publishing Company.